CLINICAL TRIAL: NCT03461757
Title: BHV3000-303: Phase 3, Double-Blind, Randomized, Placebo Controlled, Safety and Efficacy Trial of BHV-3000 (Rimegepant) Orally Disintegrating Tablet (ODT) for the Acute Treatment of Migraine
Brief Title: Trial in Adult Subjects With Acute Migraines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHV3000-303
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Results first posted 2020-03-27 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-12

CONDITIONS: Migraine, With or Without Aura
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind to Sponsor, Investigator and Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Rimegepant 75 mg (Experimental): Participants were administered a single sublingual dose of 75 mg of rimegepant ODT on occurrence of migraine that reached moderate or severe intensity up to 45 days after randomization.
  Interventions: Drug: Rimegepant
- Arm 2: Placebo (Placebo Comparator): Participants were administered a single sublingual dose of matching placebo for rimegepant (75 mg) ODT on occurrence of migraine that reached moderate or severe intensity up to 45 days after randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — 75 mg ODT QD
  Other Names: BHV-3000
  Arms: Arm 1: Rimegepant 75 mg
Drug: Placebo — Placebo ODT to match rimegepant dose QD
  Arms: Arm 2: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of BHV-3000 (rimegepant ODT) versus placebo in subjects with Acute Migraines.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject has at least 1 year history of migraines (with or without aura), consistent with a diagnosis according to the International Classification of Headache Disorder, 3rd Edition, Beta version [1] including the following:

1. Migraine attacks present for more than 1 year with the age of onset prior to 50 years of age
2. Migraine attacks, on average, lasting about 4-72 hours if untreated
3. Not more than 8 attacks of moderate to severe intensity per month within the last 3 months
4. Consistent migraine headaches of at least 2 migraine headache attacks of moderate or severe intensity in each of the 3 months prior to the Screening Visit and maintains this requirement during the Screening period
5. Less than 15 days with headache (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit and maintains this requirement during the Screening Period.
6. Subjects on prophylactic migraine medication are permitted to remain on therapy provided they have been on a stable dose for at least 3 months prior to screening visit and the dose is not expected to change during the course of the study.
7. Subjects with contraindications for use of triptans may be included provided they meet all other study entry criteria.

Key Exclusion Criteria:

1. Subject with a history of HIV disease
2. Subject history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. subjects with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening
3. Uncontrolled hypertension (high blood pressure), or uncontrolled diabetes (however subjects can be included who have stable hypertension and/or diabetes for at least 3 months prior to being enrolled)
4. Subject has a current diagnosis of major depression, other pain syndromes, psychiatric conditions (e.g., schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion might interfere with study assessments.
5. Subject has a history of gastric, or small intestinal surgery (including Gastric Bypass, Gastric Banding, Gastric Sleeve, Gastric Balloon, etc.), or has disease that causes malabsorption
6. The subject has a history of current or evidence of any significant and/ or unstable medical conditions (e.g., history of congenital heart disease or arrhythmia, known suspected infection, hepatitis B or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial.
7. History of, treatment for, or evidence of, alcohol or drug abuse within the past 12 months or subjects who have met DSM-V criteria for any significant substance use disorder within the past 12 months from the date of the screening visit.
8. Subjects are excluded if they have previously participated in any BHV-30000 (rimegepant) study within the last 2 years.
9. Participation in any other investigational clinical trial while participating in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1811 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (69):
  - Coastal Clinical Research, LLC, Mobile, Alabama
  - Clinical Research Consortium, An AMR Company, Tempe, Arizona
  - Radiant Research, Inc., Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Pharmacology Research Institute, Encino, California
  - eStudySite, La Mesa, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Synergy San Diego, National City, California
  - Pharmacology Research Institute, Newport Beach, California
  - Optimus Medical Group, San Francisco, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Yale University, New Haven, Connecticut
  - Ki Health Partners LLC DBA New England Institute for Clinical Research, Stamford, Connecticut
  - MD Clinical, Hallandale, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Qps Mra, Llc, Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Ormond Medical Arts Pharmaceutical Research, Ormond Beach, Florida
  - Synexus, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Heartland Research Associates LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Cresent City Headache and Neurology Center LLC, Chalmette, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - NECCR Primacare Research, LLC, Fall River, Massachusetts
  - Community Clinical Research Network/Milford Emergency Associates, Inc, Marlborough, Massachusetts
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Clinical Research Institute, Inc., Plymouth, Minnesota
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Hassman Research Institute, Berlin, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - CNS Research Science, Inc., Jamaica, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - PharmQuest, LLC, Greensboro, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - Radiant Research, Inc., Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Aventiv Research Inc, Dublin, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - Volunteer Research Group, Knoxville, Tennessee
  - Clinical Research Institute, Inc., Nashville, Tennessee
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Tekton Research, Inc, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Red Star Research, Lake Jackson, Texas
  - DM Clinical Research, Tomball, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin

REFERENCES:
- [Derived] Charleston L 4th, Armand CE, Monteith TS, O'Brien HL, Abbott CC, Pixton GC, Fullerton T. Efficacy and safety of rimegepant for the acute treatment of migraine in Black or African American adults: A post hoc pooled subgroup analysis from three randomized, placebo-controlled clinical trials. Headache. 2026 Feb 6. doi: 10.1111/head.70034. Online ahead of print. PMID 41652666
- [Derived] Lipton RB, Blumenfeld A, Jensen CM, Croop R, Thiry A, L'Italien G, Morris BA, Coric V, Goadsby PJ. Efficacy of rimegepant for the acute treatment of migraine based on triptan treatment experience: Pooled results from three phase 3 randomized clinical trials. Cephalalgia. 2023 Feb;43(2):3331024221141686. doi: 10.1177/03331024221141686. PMID 36739511
- [Derived] Johnston KM, Powell L, Popoff E, Harris L, Croop R, Coric V, L'Italien G. Rimegepant, Ubrogepant, and Lasmiditan in the Acute Treatment of Migraine Examining the Benefit-Risk Profile Using Number Needed to Treat/Harm. Clin J Pain. 2022 Nov 1;38(11):680-685. doi: 10.1097/AJP.0000000000001072. PMID 36125279
- [Derived] Croop R, Goadsby PJ, Stock DA, Conway CM, Forshaw M, Stock EG, Coric V, Lipton RB. Efficacy, safety, and tolerability of rimegepant orally disintegrating tablet for the acute treatment of migraine: a randomised, phase 3, double-blind, placebo-controlled trial. Lancet. 2019 Aug 31;394(10200):737-745. doi: 10.1016/S0140-6736(19)31606-X. Epub 2019 Jul 13. PMID 31311674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 69 centers in the United States.
Pre-assignment Details: Total 1811 participants were enrolled, of which 1466 were randomized to rimegepant 75 milligram (mg) orally disintegrating tablet (ODT) or placebo. Total 345 participants failed screening mainly due to failure to meet eligibility criteria. Randomization was stratified in 1:1 ratio based on use of prophylactic migraine medications (yes or no).
Groups:
- Rimegepant 75 mg ODT: Participants were administered a single sublingual dose of 75 mg of rimegepant ODT on occurrence of migraine that reached moderate or severe intensity up to 45 days after randomization.
- Placebo: Participants were administered a single sublingual dose of matching placebo for rimegepant (75 mg) ODT on occurrence of migraine that reached moderate or severe intensity up to 45 days after randomization.
Period: Overall Study
Arm/Group | Rimegepant 75 mg ODT | Placebo
Started | 732 | 734
Treated | 682 | 693
Completed | 679 | 689
Not Completed | 53 | 45
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 13 | 7
Not completed — Not Experienced Moderate/Severe Migraine | 28 | 25
Not completed — Non-compliance with study treatment | 0 | 1
Not completed — Pregnancy | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Other Reasons | 1 | 4

BASELINE CHARACTERISTICS:
Population: The analysis was performed on modified intent to treat (mITT) participants, defined as those who were randomized only once, took study medication, had moderate to severe pain level at migraine onset, and who provided at least 1 post-baseline efficacy measurement (i.e., after taking study medication).
Groups:
- Total: Total of all reporting groups
Arm/Group | Rimegepant 75 mg ODT | Placebo | Total
Number analyzed (Participants) | 669 | 682 | 1351
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.287 (12.0792) | 40.030 (11.8719) | 40.157 (11.9713)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 568 | 579 | 1147
  Male | 101 | 103 | 204
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 116 | 135 | 251
  Not Hispanic or Latino | 553 | 547 | 1100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 8 | 19 | 27
  Native Hawaiian or Other Pacific Islander | 141 | 125 | 266
  Black or African American | 11 | 5 | 16
  White | 496 | 521 | 1017
  More than one race | 7 | 9 | 16
  Unknown or Not Reported | 2 | 0 | 2
Primary Migraine Type [Count of Participants; unit: Participants]
  Migraine without Aura | 480 | 462 | 942
  Migraine with Aura | 189 | 220 | 409
Randomization Strata, Prophylactic Migraine Medication Use [Count of Participants; unit: Participants]
  Yes | 93 | 94 | 187
  No | 576 | 588 | 1164

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Pain at 2 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the electronic diary (eDiary). Pain freedom was defined as pain level of none.
Time Frame: 2 hours post-dose
Population: The analysis was performed on modified intent to treat (mITT) participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 21.2 [18.1 to 24.3] | 10.9 [8.5 to 13.2]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.4, 95% CI 2-sided [6.5 to 14.2]

2. Primary Outcome: Percentage of Participants With Freedom From Most Bothersome Symptom (MBS) at 2 Hours Post-dose
Description: MBS was reported as nausea, photophobia, or phonophobia at migraine onset using the eDiary. Symptom status (absent, present) was assessed post-dose using the eDiary separately for nausea, photophobia, and phonophobia. Freedom from MBS was defined as MBS reported at onset that was absent post-dose.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 35.1 [31.5 to 38.7] | 26.8 [23.5 to 30.2]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.3, 95% CI 2-sided [3.4 to 13.2]

3. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Pain relief was defined as pain level of none or mild.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 59.3 [55.6 to 63.1] | 43.3 [39.5 to 47.0]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.1, 95% CI 2-sided [10.8 to 21.3]

4. Secondary Outcome: Percentage of Participants With Freedom From Functional Disability at 2 Hours Post-dose
Description: Functional disability level was assessed in the eDiary on a 4-point scale: normal function, mild impairment, severe impairment, required bed rest. Freedom from functional disability was defined as normal function.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 38.1 [34.4 to 41.8] | 25.8 [22.5 to 29.1]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.1, 95% CI 2-sided [15.1 to 25.2]

5. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 24 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain relief was defined as pain level of none or mild at 2 hours up to 24 hours post-dose with no rescue medication use through 24 hours post-dose.
Time Frame: From 2 hours up to 24 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 47.8 [44.0 to 51.6] | 27.7 [24.4 to 31.1]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.1, 95% CI 2-sided [15.1 to 25.2]

6. Secondary Outcome: Percentage of Participants With Sustained Freedom From Most Bothersome Symptom (MBS) From 2 to 24 Hours Post-dose
Description: MBS was reported as nausea, photophobia, or phonophobia at migraine onset using the eDiary. Symptom status (absent, present) was assessed post-dose using the eDiary separately for nausea, photophobia, and phonophobia. Sustained freedom was defined as MBS reported at onset that was absent at 2 hours up to 24 hours post-dose with no rescue medication use through 24 hours post-dose.
Time Frame: From 2 hours up to 24 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 27.1 [23.7 to 30.4] | 17.7 [14.9 to 20.6]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.3, 95% CI 2-sided [4.9 to 13.7]

7. Secondary Outcome: Percentage of Participants With Rescue Medication Use Within 24 Hours Post-dose
Description: Participants who did not experience relief of their migraine headache at the end of 2 hours after dosing with study medication (and after the 2-hour assessments had been completed on the eDiary) were permitted to use the following rescue medications: aspirin, ibuprofen, acetaminophen up to 1000 mg/day (this includes Excedrin Migraine), naproxen (or any other type of nonsteroidal anti-inflammatory drug), antiemetics (e.g., metoclopramide or promethazine), or baclofen. The participant's use of rescue medication was recorded by the participant in a paper diary.
Time Frame: 24 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 14.2 [11.6 to 16.8] | 29.2 [25.8 to 32.6]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = -15.0, 95% CI 2-sided [-19.3 to -10.7]

8. Secondary Outcome: Percentage of Participants With Sustained Freedom From Functional Disability From 2 to 24 Hours Post-dose
Description: Functional disability level was assessed in the eDiary on a 4-point scale: normal function, mild impairment, severe impairment, required bed rest. Sustained freedom from functional disability was defined as normal function at 2 hours up to 24 hours post-dose with no rescue medication use through 24 hours post-dose.
Time Frame: From 2 hours up to 24 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 29.6 [26.1 to 33.1] | 16.9 [14.1 to 19.7]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.7, 95% CI 2-sided [8.3 to 17.2]

9. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain relief was defined as pain level of none or mild at 2 hours up to 48 hours post-dose with no rescue medication use through 48 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 42.2 [38.4 to 45.9] | 25.2 [22.0 to 28.5]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.9, 95% CI 2-sided [12.0 to 21.9]

10. Secondary Outcome: Percentage of Participants With Sustained Freedom From Most Bothersome Symptom (MBS) From 2 to 48 Hours Post-dose
Description: MBS was reported as nausea, photophobia, or phonophobia at migraine onset using the eDiary. Symptom status (absent, present) was assessed post-dose using the eDiary separately for nausea, photophobia, and phonophobia. Sustained freedom was defined as MBS reported at onset that was absent at 2 hours up to 48 hours post-dose with no rescue medication use through 48 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 23.2 [20.0 to 26.4] | 16.4 [13.6 to 19.2]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p = 0.0018, Cochran-Mantel-Haenszel; Risk Difference (RD) = 6.8, 95% CI 2-sided [2.5 to 11.0]

11. Secondary Outcome: Percentage of Participants With Sustained Freedom From Functional Disability From 2 to 48 Hours Post-dose
Description: Functional disability level was assessed in the eDiary on a 4-point scale: normal function, mild impairment, severe impairment, required bed rest. Sustained freedom from functional disability was defined as normal function at 2 hours up to 48 hours post-dose with no rescue medication use through 48 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 26.0 [22.7 to 29.3] | 15.4 [12.7 to 18.1]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.6, 95% CI 2-sided [6.3 to 14.9]

12. Secondary Outcome: Percentage of Participants With Freedom From Photophobia at 2 Hours Post-dose
Description: Photophobia (sensitivity to light) status was measured as absent or present in the eDiary. Freedom from photophobia was defined as photophobia absent.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants with photophobia present at migraine onset.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 593 | 611
percentage of participants | 33.4 [29.6 to 37.2] | 24.5 [21.1 to 28.0]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.8, 95% CI 2-sided [3.7 to 13.9]

13. Secondary Outcome: Percentage of Participants With Freedom From Functional Disability at 90 Minutes Post-dose
Description: as for outcome 4
Time Frame: 90 minutes post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 30.2 [26.7 to 33.7] | 21.3 [18.2 to 24.3]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.9, 95% CI 2-sided [4.3 to 13.6]

14. Secondary Outcome: Percentage of Participants With Pain Relief at 90 Minutes Post-dose
Description: as for outcome 3
Time Frame: 90 minutes post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 49.6 [45.8 to 53.4] | 37.2 [33.6 to 40.9]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.4, 95% CI 2-sided [7.1 to 17.6]

15. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 24 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain freedom was defined as pain level of none at 2 hours up to 24 hours post-dose with no rescue medication use through 24 hours post-dose.
Time Frame: From 2 hours up to 24 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 15.7 [12.9 to 18.4] | 5.6 [3.9 to 7.3]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.1, 95% CI 2-sided [6.9 to 13.4]

16. Secondary Outcome: Percentage of Participants With Freedom From Most Bothersome Symptom (MBS) at 90 Minutes Post-dose
Description: as for outcome 2
Time Frame: 90 minutes post dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 27.4 [24.0 to 30.7] | 21.5 [18.5 to 24.6]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p = 0.0128, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.8, 95% CI 2-sided [1.2 to 10.4]

17. Secondary Outcome: Percentage of Participants With Freedom From Pain at 90 Minutes Post-dose
Description: as for outcome 1
Time Frame: 90 minutes post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 15.1 [12.4 to 17.8] | 7.3 [5.4 to 9.3]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 7.8, 95% CI 2-sided [4.4 to 11.1]

18. Secondary Outcome: Percentage of Participants With Freedom From Phonophobia at 2 Hours Post-dose
Description: Phonophobia (sensitivity to sound) status was measured as absent or present in the eDiary. Freedom from phonophobia was defined as phonophobia absent.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants with phonophobia present at migraine onset.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 451 | 447
percentage of participants | 41.7 [37.2 to 46.3] | 30.2 [25.9 to 34.4]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.5, 95% CI 2-sided [5.3 to 17.7]

19. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain freedom was defined as pain level of none at 2 hours up to 48 hours post-dose with no rescue medication use through 48 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 13.5 [10.9 to 16.0] | 5.4 [3.7 to 7.1]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.0, 95% CI 2-sided [4.9 to 11.1]

20. Secondary Outcome: Percentage of Participants With Pain Relief at 60 Minutes Post-dose
Description: as for outcome 3
Time Frame: 60 minutes post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 36.8 [33.1 to 40.4] | 31.2 [27.8 to 34.7]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p = 0.0314, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.5, 95% CI 2-sided [0.5 to 10.6]

21. Secondary Outcome: Percentage of Participants With Freedom From Functional Disability at 60 Minutes Post-dose
Description: as for outcome 4
Time Frame: 60 minutes post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 669 | 682
percentage of participants | 22.3 [19.1 to 25.4] | 15.8 [13.1 to 18.6]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p = 0.0025, Cochran-Mantel-Haenszel; Risk Difference (RD) = 6.4, 95% CI 2-sided [2.3 to 10.6]

22. Secondary Outcome: Percentage of Participants With Freedom From Nausea at 2 Hours Post-dose
Description: Nausea status was measured as absent or present in the eDiary. Freedom from nausea was defined as nausea absent.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants with nausea present at migraine onset.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 397 | 430
percentage of participants | 51.0 [46.1 to 55.9] | 45.2 [40.5 to 49.9]
Statistical Analysis 1: Comparison: Rimegepant 75 mg ODT vs Placebo; Test type: Superiority; p = 0.0898, Cochran-Mantel-Haenszel — P-Value ≥ 0.05; therefore, all secondary endpoints listed after this endpoint in the hierarchy were not tested; Risk Difference (RD) = 5.9, 95% CI 2-sided [-0.9 to 12.7]

23. Secondary Outcome: Percentage of Participants With Pain Relapse From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Pain relapse was defined as pain level of mild, moderate, or severe after 2 hours up to 48 hours post-dose for the participants who were pain-free at 2 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The analysis population was performed on mITT participants with pain freedom at 2 hours post-dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rimegepant 75 mg ODT | Placebo
Number analyzed (Participants) | 142 | 74
percentage of participants | 36.6 [28.7 to 44.5] | 50.0 [38.7 to 61.2]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected from informed consent up to the end of the study, and adverse events (AEs) were collected from randomization up to end of the study (up to 52 days).
Description: The safety population, all enrolled participants who received at least 1 dose of rimegepant or placebo, was used to determine the number of participants at risk for SAEs and Other AEs.
Arm/Group | Rimegepant 75 mg ODT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/682 | 0/693
Serious Adverse Events (participants affected / at risk) | 0/682 | 0/693
Other Adverse Events (participants affected / at risk) | 0/682 | 0/693

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03461757/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT03461757/SAP_001.pdf